CLINICAL TRIAL: NCT02343939
Title: A Phase 1b/2 Study of Entospletinib (GS-9973) Monotherapy and in Combination With Chemotherapy in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Entospletinib Monotherapy and in Combination With Chemotherapy in Adults With Acute Myeloid Leukemia (AML)
Acronym: ENTO in AML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-1559; 2016-003353-16 (EudraCT Number)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Daunorubicin; Cytarabine; Decitabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Entospletinib + daunorubicin + cytarabine (Group A) (Experimental): Dose Escalation: Entospletinib up to 400 mg for 14 days and then entospletinib up to 400 mg in combination with daunorubicin and cytarabine for up to two 14-day cycles.
  Dose Expansion: Entospletinib 400 mg for 14 days and then entospletinib 400 mg in combination with daunorubicin and cytarabine for up to two 14-day cycles. Some participants will have the option to receive post-induction therapy with entospletinib 400 mg in combination with cytarabine/cytosine arabinoside (ARA-C). Participants may receive maintenance therapy with 28-day cycles of entospletinib 400 mg for up to twelve 28-day cycles, if the participant is not eligible for stem cell transplant.
  Interventions: Drug: Entospletinib; Drug: Daunorubicin; Drug: Cytarabine
- Entospletinib + decitabine (Group B) (Experimental): Dose Escalation: Entospletinib 400 mg for 14 days and then entospletinib 400 mg in combination with decitabine for 10 days beginning on Day 1 of every 28-day cycle (at least 2 cycles of induction therapy but no more than 4 cycles). Participants who are intolerant of decitabine may switch to entospletinib monotherapy maintenance at any time after completing the first 2 cycles.
  Dose Expansion: Entospletinib 400 mg for 14 days for the safety run-in participants or Entospletinib 400 mg for 5 days for the randomization participants. Then entospletinib 400 mg in combination with decitabine or azacitidine (at least 2 cycles of induction therapy but no more than 4 cycles). Some participants will have the option to receive maintenance therapy with entospletinib in combination with decitabine or azacitidine. Participants who are intolerant of decitabine or azacitidine may switch to entospletinib monotherapy maintenance at any time after completing the first 2 cycles.
  Interventions: Drug: Entospletinib; Drug: Decitabine; Drug: Azacitidine
- Entospletinib (Group C) (Experimental): Dose Escalation: Entospletinib up to 800 mg for 28-day cycles until the participant meets criteria for study treatment discontinuation per the study protocol.
  Dose Expansion: Entospletinib 400 mg for 28-day cycles until the participant meets criteria for study treatment discontinuation per the protocol.
  Interventions: Drug: Entospletinib

INTERVENTIONS:
Drug: Entospletinib — Tablet(s) administered orally every 12 hours
  Other Names: GS-9973; ENTO
Drug: Daunorubicin — 60 mg/m^2 administered intravenously daily on Days 1 to 3 for up to two 14-day induction cycles
  Arms: Entospletinib + daunorubicin + cytarabine (Group A)
Drug: Cytarabine — 100 mg/m^2 administered intravenously daily on Days 1 to 7 for up to two 14-day cycles
  Arms: Entospletinib + daunorubicin + cytarabine (Group A)
Drug: Decitabine — 20 mg/m^2 administered intravenously
  Arms: Entospletinib + decitabine (Group B)
Drug: Azacitidine — 75 mg/m^2 administered intravenously or subcutaneously
  Arms: Entospletinib + decitabine (Group B)

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of entospletinib when administered as monotherapy or in combination with chemotherapy in adults with acute myeloid leukemia (AML).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with AML in need of treatment
* Group A : Individuals ≥ 18 years of age with previously untreated AML by World Health Organization (WHO) criteria who are able and should receive up to 2 cycles of induction chemotherapy with 7+3 as determined by the treating physician
* Group B: Individuals > 70 years of age with previously untreated AML by WHO criteria; or individuals ≤ 70 years of age with previously untreated AML who refuse or are unable to receive chemotherapy with 7+3 as determined by the treating physician
* Group C: Individuals ≥ 18 years of age with relapsed/refractory AML by WHO criteria; or with relapsed/refractory AML with mixed-lineage leukemia (MLL); or with previously untreated AML by WHO criteria and who would have met disease eligibility criteria for Group A or B but refuse or are unable to receive chemotherapy and hypomethylating agent as determined by the treating physician

Key Exclusion Criteria:

* Known active central nervous system or leptomeningeal lymphoma
* Subjects with acute promyelocytic leukemia (M3)
* Treatment with proton pump inhibitors (PPIs) within 7 days prior to enrollment.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (17):
- United States (14):
  - UCLA, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc, Fairway, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medical College - New York - Presbyterian Hospital, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Saint Francis Cancer Center, Greenville, South Carolina
- Canada (2):
  - Princess Margaret, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Universitätsklinikum Frankfurt Medizinische Klinik II, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, Canada, and Germany. The first participant was screened on 01 July 2015.
Pre-assignment Details: 233 participants were screened.
Groups:
- Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin: Participants received ENTO 200 mg tablet orally every 12 hours on Days 1 to 14 (Cycle 0) (during monotherapy lead-in), followed by ENTO 200 mg tablet orally every 12 hours in combination with chemotherapy (cytarabine 100 mg/m^2 on Days 1-7 and daunorubicin 60 mg/m^2 on Days 1-3 intravenously) for up to two 14-day cycles (Cycles 1 and 2) (during induction chemotherapy).
- Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin: Phase1b/2: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1 to 14 (Cycle 0) (monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with chemotherapy (cytarabine 100 mg/m^2 on Days 1-7 and daunorubicin 60 mg/m^2 on Days 1-3 intravenously) for up to two 14-day cycles (Cycles 1 and 2) (induction chemotherapy).
  Phase 2 only: Participants who achieved a CR/CRi and did not require or could not proceed to allogeneic stem cell transplantation (SCT) were offered post-remission chemotherapy (cytarabine 3 g/m^2 intravenously every 12 hours on Days 1, 3, and 5 or 1 g/m^2 intravenously once daily on Days 1-5) in combination with ENTO 400 mg tablet orally every 12 hours on Days 1-28 of each 28-day cycle for at least 3 and up to 4 cycles. Participants who maintained a CR/CRi after 3 or 4 cycles were offered maintenance therapy with ENTO 400 mg tablet orally every 12 hours on Days 1-28 of each 28-day cycle for up to 12 cycles.
- Group B Phase 1b ENTO 200 mg + Decitabine: Participants received ENTO 200 mg tablet orally every 12 hours on Days 1-14 (Cycle 0) (during monotherapy lead-in), followed by ENTO 200 mg tablet orally every 12 hours in combination with decitabine 20 mg/m^2 intravenously on Days 1-10 of every 28-day cycle for 2 cycles (or up to 4 cycles for participants with persistent disease after Cycle 2 Day 28) (induction chemotherapy). Participants who achieved a CR/CRi received SCT (if eligible) per investigator's discretion; other participants were offered maintenance therapy with ENTO every 12 hours on Days 1-28 in combination with decitabine on Days 1-5 of every 28-day cycle for at least 2 cycles (maximum up to 12 cycles). Participants who were intolerant to decitabine were offered maintenance therapy with ENTO 200 mg as monotherapy after completing 2 maintenance cycles.
- Group B Phase 1b ENTO 400 mg + Decitabine: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1-14 (Cycle 0) (during monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with decitabine 20 mg/m^2 intravenously on Days 1-10 of every 28-day cycle for 2 cycles (or up to 4 cycles for participants with persistent disease after Cycle 2 Day 28) (induction chemotherapy). Participants who achieved a CR/CRi received SCT (if eligible) per investigator's discretion; other participants were offered maintenance therapy with ENTO every 12 hours on Days 1-28 in combination with decitabine on Days 1-5 of every 28-day cycle for at least 2 cycles (maximum up to 12 cycles). Participants who were intolerant to decitabine were offered maintenance therapy with ENTO 400 mg as monotherapy after completing 2 maintenance cycles.
- Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In): As part of the safety run-in, participants received ENTO 400 mg tablet orally every 12 hours on Days 1-14 (Cycle 0) (during monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with azacitidine 75 mg/m^2 intravenously on Days 1-7 of a 28-day cycle (Cycle 1). Participants who were not eligible for SCT were offered maintenance therapy with ENTO every 12 hours on Days 1-28 in combination with azacitidine on Days 1-7 of every 28-day cycle for at least 2 cycles (maximum up to 12 cycles). Participants who were intolerant to azacitidine were offered maintenance therapy with ENTO 400 mg as monotherapy after completing 2 maintenance cycles.
- Group B Phase 2 ENTO 400 mg + Decitabine (Randomized): Participants were randomized to receive ENTO 400 mg tablet orally every 12 hours on Days 1-5 (Cycle 0) (during monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with decitabine 20 mg/m^2 intravenously on Days 1-10 of every 28-day cycle for 2 cycles (or up to 4 cycles for participants with persistent disease after Cycle 2 Day 28). Participants who were not eligible for SCT were offered maintenance therapy with ENTO every 12 hours on Days 1-28 in combination with decitabine on Days 1-5 of every 28-day cycle for at least 2 cycles (maximum up to 12 cycles). Participants who were intolerant to decitabine were offered maintenance therapy with ENTO 400 mg as monotherapy after completing 2 maintenance cycles.
- Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized): Participants were randomized to receive ENTO 400 mg tablet orally every 12 hours on Days 1-5 (Cycle 0) (during monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with azacitidine 75 mg/m^2 intravenously on Days 1-7 of every 28-day cycle for 2 cycles (or up to 4 cycles for participants with persistent disease after Cycle 2 Day 28). Participants who were not eligible for SCT were offered maintenance therapy with ENTO every 12 hours on Days 1-28 in combination with azacitidine on Days 1-7 of every 28-day cycle for at least 2 cycles (maximum up to 12 cycles). Participants who were intolerant to azacitidine were offered maintenance therapy with ENTO 400 mg as monotherapy after completing 2 maintenance cycles.
- Group C Phase 1b/2 ENTO 400 mg: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
- Group C Phase 1b ENTO 800 mg: Participants received ENTO 800 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
Period: Overall Study
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
Started | 3 | 50 | 5 | 6 | 8 | 17 | 15 | 37 | 7
Completed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 48 | 5 | 6 | 8 | 17 | 15 | 37 | 7
Not completed — Death | 0 | 15 | 4 | 2 | 5 | 11 | 8 | 22 | 1
Not completed — Study terminated by sponsor | 0 | 27 | 0 | 1 | 1 | 5 | 3 | 4 | 0
Not completed — Withdrew consent | 3 | 6 | 1 | 2 | 2 | 0 | 0 | 8 | 6
Not completed — Treatment failure | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Investigator's discretion | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Never Treated With ENTO | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received at least 1 dose of study drug with treatment designated according to the planned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Total
Number analyzed (Participants) | 3 | 50 | 5 | 6 | 8 | 17 | 14 | 35 | 7 | 145
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 3 | 32 | 0 | 1 | 1 | 1 | 0 | 17 | 0 | 55
  ≥ 65 years | 0 | 18 | 5 | 5 | 7 | 16 | 14 | 18 | 7 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 21 | 2 | 2 | 2 | 7 | 3 | 18 | 5 | 61
  Male | 2 | 29 | 3 | 4 | 6 | 10 | 11 | 17 | 2 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
  Ethnicity: Not Hispanic or Latino | 3 | 48 | 5 | 6 | 7 | 15 | 13 | 33 | 7 | 137
  Ethnicity: Not Permitted | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 3 | 44 | 3 | 6 | 6 | 14 | 11 | 31 | 7 | 125
  Race: Black or African American | 0 | 5 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 11
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Other | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Race: Not Permitted | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 10
  United States | 3 | 46 | 5 | 6 | 8 | 15 | 11 | 29 | 7 | 130
  Germany | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: DLTs refer to toxicities experienced during the first 28 days of study treatment that have been judged to be clinically significant and related to study treatment. DLT assessment was applicable only for Phase 1b and Phase 2 safety run-in participants.
Time Frame: Group A: Cycle 0 Day 1 to Cycle 2 Day 28; Group B: Cycle 0 Day 1 to Cycle 1 Day 28; Group C: Cycle 1 Day 1 to Cycle 1 Day 28 (Cycle length: for Cycle 0 = 14 days, for all other cycles = 28 days)
Population: The DLT Analysis Set included all participants who received 21 days of ENTO (applicable to all groups) and all doses of cytarabine and daunorubicin in Group A Phase 1b, decitabine in Group B Phase 1b, or azacitidine in Group B Phase 2 safety run-in during the DLT assessment window; or experienced a DLT during the DLT assessment window.
Measure: Number; unit: percentage of participants
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 16.7 | 0 | 0 | 16.7

2. Primary Outcome: Percentage of Participants With Morphologic Complete Remission (CR) at the End of Induction
Description: Clinical response was assessed according to the International Working Group criteria (Cheson 2003). Morphologic CR included CR and cytogenetic CR (CRc). CR required all of the following: < 5% blasts in bone marrow aspirate; Neutrophils ≥ 1,000/microliter (mcL); Platelets ≥ 100,000/mcL; No extramedullary disease; No blasts with Auer rods detected; and Independent of transfusions. CRc, in addition to CR criteria, required reversion to a normal karyotype with an abnormal karyotype at the time of diagnosis.
Time Frame: At the end of induction (Group A: up to end of Cycle 2; Group B: up to end of Cycle 4) (cycle length = up to 28 days); Group C: From Day 1 until meeting the criteria for study treatment discontinuation (up to approximately 3 years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1 to 14 (Cycle 0) (during monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with chemotherapy (cytarabine 100 mg/m^2 on Days 1-7 and daunorubicin 60 mg/m^2 on Days 1-3 intravenously) for up to two 14-day cycles (Cycles 1 and 2) (during induction chemotherapy).
- Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1-14 (Cycle 0) (monotherapy lead-in), followed by ENTO 400 mg tablet orally every 12 hours in combination with chemotherapy (cytarabine 100 mg/m^2 on Days 1-7 and daunorubicin 60 mg/m^2 on Days 1-3 intravenously) for up to two 14-day cycles (Cycles 1 and 2) (induction chemotherapy). Participants who achieved a CR/CRi and did not require or could not proceed to allogeneic stem cell transplantation (SCT) were offered post-remission chemotherapy (cytarabine 3 g/m^2 intravenously every 12 hours on Days 1, 3, and 5 or 1 g/m^2 intravenously once daily on Days 1-5) in combination with ENTO 400 mg tablet orally every 12 hours on Days 1-28 of each 28-day cycle for at least 3 and up to 4 cycles. Participants who maintained a CR/CRi after 3 or 4 cycles were offered maintenance therapy with ENTO 400 mg tablet orally every 12 hours on Days 1-28 of each 28-day cycle for up to 12 cycles.
- Group C Phase 1b ENTO 400 mg: Participants received ENTO 400 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
- Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML): Participants with relapsed/refractory (R/R) acute myeloid leukemia (AML) received ENTO 400 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
- Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL): Participants R/R AML with mixed-lineage leukemia (MLL) received ENTO 400 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
- Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML): Participants with previously untreated AML who were unfit for chemotherapy or hypomethylating agents or refused chemotherapy or hypomethylating agent received ENTO 400 mg tablet orally every 12 hours on Days 1-28 of every 28-day cycle until treatment failure, start of new therapy, unacceptable toxicity, withdrawal of consent, withdrawal from study by investigator, or study termination by sponsor.
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin | Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML) | Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL) | Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML)
Number analyzed (Participants) | 3 | 9 | 41 | 5 | 6 | 8 | 17 | 14 | 7 | 7 | 6 | 13 | 9
percentage of participants | 66.7 [9.4 to 99.2] | 66.7 [29.9 to 92.5] | 46.3 [30.7 to 62.6] | 0.0 [0.0 to 52.2] | 16.7 [0.4 to 64.1] | 25.0 [3.2 to 65.1] | 0.0 [0.0 to 19.5] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 15.4 [1.9 to 45.4] | 11.1 [0.3 to 48.2]

3. Primary Outcome: Percentage of Participants With Composite Complete Remission at the End of Induction
Description: Clinical response was assessed according to the International Working Group criteria (Cheson 2003). Composite complete remission included CR, CRc, and morphologic complete remission with incomplete blood count recovery (CRi). CR required all of the following: < 5% blasts in bone marrow aspirate; Neutrophils ≥ 1,000/mcL; Platelets ≥ 100,000/mcL; No extramedullary disease; No blasts with Auer rods detected; and Independent of transfusions. CRc, in addition to CR criteria, required reversion to a normal karyotype with an abnormal karyotype at the time of diagnosis. CRi required all of the CR criteria except the criterion of neutrophils and platelets.
Time Frame: as for outcome 2
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin | Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML) | Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL) | Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML)
Number analyzed (Participants) | 3 | 9 | 41 | 5 | 6 | 8 | 17 | 14 | 7 | 7 | 6 | 13 | 9
percentage of participants | 100.0 [29.2 to 100] | 77.8 [40 to 97.2] | 65.9 [49.4 to 79.9] | 40.0 [5.3 to 85.3] | 50.0 [11.8 to 88.2] | 25.0 [3.2 to 65.1] | 23.5 [6.8 to 49.9] | 14.3 [1.8 to 42.8] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 15.4 [1.9 to 45.4] | 11.1 [0.3 to 48.2]

4. Primary Outcome: Percentage of Participants With Overall Response at the End of Induction
Description: Clinical response was assessed according to the International Working Group criteria (Cheson 2003). Overall response included CR, CRc, CRi, and partial remission (PR). CR required all of the following: < 5% blasts in bone marrow aspirate; Neutrophils ≥ 1,000/mcL; Platelets ≥ 100,000/mcL; No extramedullary disease; No blasts with Auer rods detected; and Independent of transfusions. CRc, in addition to CR criteria, required reversion to a normal karyotype with an abnormal karyotype at the time of diagnosis. CRi required all of the CR criteria except the criterion of neutrophils and platelets. PR required all of the following: ≥ 50% decrease in blasts in bone marrow aspirate to a range of 5% to 25%; Neutrophils ≥ 1,000/mcL; Platelets ≥ 100,000/mcL; Independent of transfusions; and A value of ≤ 5% blasts was also considered a PR if Auer rods were detected.
Time Frame: as for outcome 2
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin | Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML) | Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL) | Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML)
Number analyzed (Participants) | 3 | 9 | 41 | 5 | 6 | 8 | 17 | 14 | 7 | 7 | 6 | 13 | 9
percentage of participants | 100.0 [29.2 to 100] | 77.8 [40 to 97.2] | 70.7 [54.5 to 83.9] | 40.0 [5.3 to 85.3] | 50.0 [11.8 to 88.2] | 25.0 [3.2 to 65.1] | 23.5 [6.8 to 49.9] | 14.3 [1.8 to 42.8] | 14.3 [0.4 to 57.9] | 0.0 [0 to 41] | 0.0 [0 to 45.9] | 15.4 [1.9 to 45.4] | 11.1 [0.3 to 48.2]

5. Secondary Outcome: Duration of Exposure of Entospletinib
Time Frame: First dose date up to approximately 3 years
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: weeks
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
Number analyzed (Participants) | 3 | 50 | 5 | 6 | 8 | 17 | 14 | 35 | 7
weeks | 8.6 [6.1 to 10.0] | 7.1 [0.9 to 72.9] | 13.7 [1.6 to 50.9] | 15.4 [1.9 to 58.9] | 10.1 [1.3 to 39.4] | 13.9 [1.9 to 40.0] | 10.1 [0.9 to 47.0] | 4.4 [1.4 to 15.6] | 7.6 [2.0 to 9.0]

6. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time interval from the start of the study therapy until the date of treatment failure, acute myeloid leukemia (AML) relapse, or death from any cause, whichever occurred first. Participants who received other anti-cancer therapy (prior to the event if any) were censored. Median EFS was analyzed using Kaplan-Meier (KM) method.
Time Frame: First dose date up to approximately 38 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin | Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML) | Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL) | Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML)
Number analyzed (Participants) | 3 | 9 | 41 | 5 | 6 | 8 | 17 | 14 | 7 | 7 | 6 | 13 | 9
months | NA [NA to NA] — Median and confidence interval limits could not be calculated due to low number of participants with an event. | 1.9 [0.9 to 1.9] | 9.0 [2.3 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | 2.2 [0.5 to 4.7] | 2.9 [1.1 to 7.7] | 2.3 [0.5 to 9.0] | 3.2 [0.5 to 4.2] | 2.4 [2.1 to 3.9] | 1.8 [0.9 to 1.9] | 1.8 [0.5 to 1.9] | 1.0 [0.7 to 2.8] | 1.0 [0.8 to 2.7] | 1.7 [0.8 to 1.9]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the start of the study therapy to death from any cause. Median OS was analyzed using KM method.
Time Frame: First dose date up to approximately 38 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b ENTO 400 mg + Cytarabine + Daunorubicin | Group A Phase 2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b ENTO 400 mg | Group C Phase 1b ENTO 800 mg | Group C Phase 2 ENTO 400 mg (Cohort C1A - R/R AML) | Group C Phase 2 ENTO 400 mg (Cohort C2 - MLL) | Group C Phase 2 ENTO 400 mg (Cohort C3 - Untreated AML)
Number analyzed (Participants) | 3 | 9 | 41 | 5 | 6 | 8 | 17 | 14 | 7 | 7 | 6 | 13 | 9
months | 37.1 [9.1 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | 34.1 [1.2 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | NA [16.8 to NA] — Median and upper limit of confidence interval could not be calculated due to low number of participants with an event. | 3.2 [0.8 to 12.7] | 5.3 [2.4 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | 6.9 [1.4 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | 7.3 [2.4 to NA] — Upper limit of confidence interval could not be calculated due to low number of participants with an event. | 6.2 [3.2 to 10.2] | 5.9 [0.9 to 6.3] | 5.6 [0.5 to 8.4] | 8.2 [0.7 to 24.3] | 7.9 [3.3 to 11.9] | 2.2 [1.0 to 4.7]

8. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 18 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
Number analyzed (Participants) | 3 | 50 | 5 | 6 | 8 | 17 | 14 | 35 | 7
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

9. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 18 months)
Population: Participants in the Safety Analysis Set who had non-missing postbaseline value prior to or on the last dosing date plus 30 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
Number analyzed (Participants) | 3 | 50 | 5 | 6 | 7 | 17 | 14 | 35 | 7
percentage of participants
  Any Laboratory Abnormality | 100 | 100 | 100 | 100 | 100 | 94.1 | 100 | 100 | 100
  Grade 3 or 4 Laboratory Abnormalities | 100 | 98.0 | 100 | 100 | 85.7 | 94.1 | 92.9 | 82.9 | 85.7

ADVERSE EVENTS:
Time Frame: - All-Cause Mortality: First dose date up to approximately 38 months. - Adverse Events: First dose date up to the last dose date plus 30 days (maximum: 18 months)
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin | Group B Phase 1b ENTO 200 mg + Decitabine | Group B Phase 1b ENTO 400 mg + Decitabine | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) | Group C Phase 1b/2 ENTO 400 mg | Group C Phase 1b ENTO 800 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 21/50 | 5/5 | 4/6 | 5/8 | 12/17 | 11/14 | 30/35 | 6/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 23/50 | 5/5 | 5/6 | 7/8 | 11/17 | 7/14 | 19/35 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 50/50 | 5/5 | 6/6 | 7/8 | 17/17 | 14/14 | 33/35 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin (N=3) | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin (N=50) | Group B Phase 1b ENTO 200 mg + Decitabine (N=5) | Group B Phase 1b ENTO 400 mg + Decitabine (N=6) | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) (N=8) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) (N=17) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) (N=14) | Group C Phase 1b/2 ENTO 400 mg (N=35) | Group C Phase 1b ENTO 800 mg (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 13 | 4 | 4 | 3 | 8 | 0 | 5 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Phase 1b ENTO 200 mg + Cytarabine + Daunorubicin (N=3) | Group A Phase 1b/2 ENTO 400 mg + Cytarabine + Daunorubicin (N=50) | Group B Phase 1b ENTO 200 mg + Decitabine (N=5) | Group B Phase 1b ENTO 400 mg + Decitabine (N=6) | Group B Phase 2 ENTO 400 mg + Azacitidine (Safety Run-In) (N=8) | Group B Phase 2 ENTO 400 mg + Decitabine (Randomized) (N=17) | Group B Phase 2 ENTO 400 mg + Azacitidine (Randomized) (N=14) | Group C Phase 1b/2 ENTO 400 mg (N=35) | Group C Phase 1b ENTO 800 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 24 | 3 | 1 | 2 | 5 | 6 | 10 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 36 | 1 | 3 | 2 | 2 | 4 | 8 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 7 | 1 | 0 | 1 | 3 | 3 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 6 | 0 | 2 | 1 | 2 | 2 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve cupping (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scleral hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 10 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 7 | 0 | 2 | 0 | 0 | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 13 | 0 | 1 | 0 | 1 | 4 | 4 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 20 | 3 | 4 | 6 | 10 | 9 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 34 | 1 | 3 | 3 | 9 | 4 | 14 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 8 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 6 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 5 | 0 | 1 | 0 | 3 | 1 | 3 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 34 | 4 | 4 | 4 | 5 | 7 | 15 | 2
Oral pain (Gastrointestinal disorders) | 0 | 5 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 8 | 1 | 1 | 0 | 4 | 1 | 6 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 16 | 0 | 1 | 1 | 6 | 5 | 8 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Catheter site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Chills (General disorders) | 0 | 8 | 0 | 0 | 0 | 2 | 5 | 4 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 14 | 3 | 1 | 2 | 9 | 6 | 10 | 3
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 10 | 1 | 0 | 0 | 0 | 1 | 4 | 0
Non-cardiac chest pain (General disorders) | 0 | 7 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 29 | 2 | 3 | 4 | 6 | 4 | 4 | 3
Pain (General disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 9 | 0 | 2 | 2 | 2 | 1 | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 9 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Leptotrichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 11 | 1 | 2 | 1 | 1 | 0 | 3 | 0
Mucosal infection (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 1 | 1 | 3 | 0 | 3 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 4 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 6 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 8 | 0 | 0 | 2 | 0 | 1 | 4 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 8 | 0 | 0 | 2 | 1 | 2 | 3 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 12 | 0 | 0 | 2 | 5 | 4 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 6 | 1 | 1 | 1 | 1 | 7 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 5 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 1 | 1 | 2 | 4 | 0 | 1 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 16 | 2 | 2 | 2 | 4 | 2 | 6 | 2
Platelet count decreased (Investigations) | 0 | 26 | 3 | 3 | 3 | 5 | 7 | 9 | 1
Spleen palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ultrasound liver abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 3 | 2 | 1 | 0
Weight increased (Investigations) | 2 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 18 | 2 | 1 | 2 | 7 | 5 | 4 | 1
White blood cell count increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 22 | 2 | 1 | 3 | 6 | 6 | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 10 | 1 | 0 | 1 | 3 | 3 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 7 | 1 | 0 | 1 | 2 | 4 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1 | 0 | 4 | 5 | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 2 | 4 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1 | 0 | 0 | 2 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0 | 2 | 0 | 1 | 0 | 6 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 2 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 4 | 1 | 3 | 1
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 14 | 0 | 0 | 0 | 1 | 1 | 5 | 0
Dysgeusia (Nervous system disorders) | 0 | 11 | 0 | 1 | 3 | 2 | 3 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 20 | 2 | 3 | 0 | 3 | 2 | 6 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 7 | 1 | 2 | 0 | 1 | 0 | 3 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 5 | 1 | 0 | 1 | 2 | 0 | 2 | 1
Delirium (Psychiatric disorders) | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 16 | 2 | 1 | 1 | 2 | 4 | 7 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 8 | 0 | 0 | 1 | 2 | 3 | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 5 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 18 | 1 | 4 | 3 | 5 | 5 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 20 | 2 | 3 | 2 | 5 | 4 | 10 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 1 | 2 | 0 | 3 | 2 | 7 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 1 | 1 | 0 | 2 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 0 | 0 | 0 | 3 | 1 | 2 | 0
Paranasal sinus hyposecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0 | 3 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 6 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 0 | 2 | 2 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 21 | 1 | 3 | 0 | 0 | 1 | 8 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 12 | 0 | 3 | 0 | 3 | 0 | 2 | 1
Hypotension (Vascular disorders) | 1 | 7 | 0 | 0 | 2 | 4 | 5 | 6 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT02343939/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT02343939/SAP_001.pdf